CLINICAL TRIAL: NCT04805073
Title: Assessing Efficacy of Intramuscular Promethazine for the Treatment of Intrathecal Morphine Induced Pruritus
Brief Title: Treatment of Pruritus With Intramuscular Promethazine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB202002297-A; OCR40099 (Other: UFOnCore)
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Pruritus; Pregnancy Related
Keywords: cesarean section
MeSH Terms: conditions — Pruritus | interventions — Promethazine; Fluoridation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Stratified randomization design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Promethazine (Experimental): The treatment will consist of a blinded syringe of 1cc clear liquid 25mg/ml Promethazine
  Interventions: Drug: Promethazine
- Placebo (Placebo Comparator): The treatment will consist of a blinded syringe of 1cc 0.9% Sodium Chloride
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Promethazine — 1cc 25mg/ml Promethazine (study medication)
  Other Names: Phenergan
  Arms: Promethazine
Drug: Placebo — 1cc 0.9% Sodium Chloride (placebo)
  Other Names: salt water
  Arms: Placebo

SUMMARY:
Neuraxial narcotics are commonly used in obstetric patients for cesarean delivery to help with pain control over the first 24 hours after the surgery. The aim is to evaluate effectiveness of promethazine (IMP) treatment of intrathecal morphine induced pruritus (ITIMIP). A treatment for ITMIP, other than naloxone, will allow for increased use of intrathecal narcotics and decrease the use of systemic opioids in the initial post-operative period.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant adult female patients of at least 18 years of age consenting to a cesarean birth
* Willing to consent to study.

Exclusion Criteria:

* Male patients
* Incarceration
* Inability to communicate with the investigators
* Allergies to any medications used in the study
* Possessing any contraindication to spinal anesthesia (lack of consent, elevated intracranial pressure, preexisting neurological disease, thrombocytopenia/coagulopathy, hypovolemia, infection at the site of the procedure)
* Patients with an already prolonged QTc (>500 ms)
* Any reason an investigator believes study participation would not be in the best interest of the potential subject.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant adult female patients of at least 18 years of age consenting to a cesarean birth.
Enrollment: 72 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Wendling, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morgan PJ, Mehta S, Kapala DM. Nalbuphine pretreatment in cesarean section patients receiving epidural morphine. Reg Anesth. 1991 Mar-Apr;16(2):84-8. PMID 2043531
- [Background] Cohen SE, Ratner EF, Kreitzman TR, Archer JH, Mignano LR. Nalbuphine is better than naloxone for treatment of side effects after epidural morphine. Anesth Analg. 1992 Nov;75(5):747-52. PMID 1416128
- [Background] Vice-O'Con K, Austin PN, Pugh MA. Pharmacologic Methods for Preventing Pruritus in Patients Receiving Intrathecal Opioids for Cesarean Delivery. AANA J. 2018 Feb;86(1):59-66. PMID 31573495
- [Background] Penning JP, Samson B, Baxter AD. Reversal of epidural morphine-induced respiratory depression and pruritus with nalbuphine. Can J Anaesth. 1988 Nov;35(6):599-604. doi: 10.1007/BF03020347. PMID 3144443
- [Background] Alhashemi JA, Crosby ET, Grodecki W, Duffy PJ, Hull KA, Gallant C. Treatment of intrathecal morphine-induced pruritus following caesarean section. Can J Anaesth. 1997 Oct;44(10):1060-5. doi: 10.1007/BF03019227. PMID 9350364
- [Background] Ituk U, Habib AS. Enhanced recovery after cesarean delivery. F1000Res. 2018 Apr 27;7:F1000 Faculty Rev-513. doi: 10.12688/f1000research.13895.1. eCollection 2018. PMID 29770203
- [Background] Singh PM, Sultan P, O'Carroll J, Blake L, Carvalho B, Singh NP, Monks DT. Pharmacological agents for prevention of pruritus in women undergoing Caesarean delivery with neuraxial morphine: a systematic review and Bayesian network meta-analysis. Br J Anaesth. 2023 Sep;131(3):556-571. doi: 10.1016/j.bja.2023.05.028. Epub 2023 Jul 14. PMID 37455197
- [Background] Moustafa AA, Baaror AS, Abdelazim IA. Comparative study between nalbuphine and ondansetron in prevention of intrathecal morphine-induced pruritus in women undergoing cesarean section. Anesth Essays Res. 2016 May-Aug;10(2):238-44. doi: 10.4103/0259-1162.167839. PMID 27212754
- [Background] Charuluxananan S, Somboonviboon W, Kyokong O, Nimcharoendee K. Ondansetron for treatment of intrathecal morphine-induced pruritus after cesarean delivery. Reg Anesth Pain Med. 2000 Sep-Oct;25(5):535-9. doi: 10.1053/rapm.2000.7809. PMID 11009242
- [Background] Sultan P, Halpern SH, Pushpanathan E, Patel S, Carvalho B. The Effect of Intrathecal Morphine Dose on Outcomes After Elective Cesarean Delivery: A Meta-Analysis. Anesth Analg. 2016 Jul;123(1):154-64. doi: 10.1213/ANE.0000000000001255. PMID 27089000
- [Background] Kumar K, Singh SI. Neuraxial opioid-induced pruritus: An update. J Anaesthesiol Clin Pharmacol. 2013 Jul;29(3):303-7. doi: 10.4103/0970-9185.117045. PMID 24106351
- [Background] Ito S, Blajchman A, Stephenson M, Eliopoulos C, Koren G. Prospective follow-up of adverse reactions in breast-fed infants exposed to maternal medication. Am J Obstet Gynecol. 1993 May;168(5):1393-9. doi: 10.1016/s0002-9378(11)90771-6. PMID 8498418
- [Background] Anwari JS, Iqbal S. Antihistamines and potentiation of opioid induced sedation and respiratory depression. Anaesthesia. 2003 May;58(5):494-5. doi: 10.1046/j.1365-2044.2003.03154_18.x. No abstract available. PMID 12694022
- [Result] Eldor J, Fishelev V, Levine S, Guedj P, Dudakova I. Prevention of epidural morphine pruritus by intramuscular promethazine in parturients. Reg Anesth. 1994 Nov-Dec;19(6):433-4. No abstract available. PMID 7848959
- [Result] Slappendel R, Weber EW, Benraad B, van Limbeek J, Dirksen R. Itching after intrathecal morphine. Incidence and treatment. Eur J Anaesthesiol. 2000 Oct;17(10):616-21. doi: 10.1046/j.1365-2346.2000.00727.x. PMID 11050519
- [Result] Horta ML, Morejon LC, da Cruz AW, Dos Santos GR, Welling LC, Terhorst L, Costa RC, Alam RU. Study of the prophylactic effect of droperidol, alizapride, propofol and promethazine on spinal morphine-induced pruritus. Br J Anaesth. 2006 Jun;96(6):796-800. doi: 10.1093/bja/ael072. Epub 2006 Apr 5. PMID 16597655
- [Result] Haydek CG, Love E, Mollanazar NK, Valdes Rodriguez R, Lee H, Yosipovitch G, Tharp MD, Hanifin JM, Chen KH, Chen SC. Validation and Banding of the ItchyQuant: A Self-Report Itch Severity Scale. J Invest Dermatol. 2017 Jan;137(1):57-61. doi: 10.1016/j.jid.2016.06.633. Epub 2016 Aug 10. PMID 27521593
- [Result] Koju RB, Gurung BS, Dongol Y. Prophylactic administration of ondansetron in prevention of intrathecal morphine-induced pruritus and post-operative nausea and vomiting in patients undergoing caesarean section. BMC Anesthesiol. 2015 Feb 17;15:18. doi: 10.1186/1471-2253-15-18. PMID 25971957

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Promethazine | Placebo
Started | 36 | 36
Completed | 34 | 33
Not Completed | 2 | 3
Not completed — study personnel not available | 2 | 0
Not completed — spinal anesthesia failure | 0 | 1
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: Not recorded
Groups:
- Total: Total of all reporting groups
Arm/Group | Promethazine | Placebo | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 36 | 72
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 36 | 72
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 36 | 36 | 72

OUTCOME MEASURES:

1. Primary Outcome: Does the Addition of Promethazine Reduce Itching After Spinal Morphine for Cesarean Delivery?
Description: Pruritus (itching) will be quantified by the ItchyQuant Scale. The ItchyQuant scale is a 0 -10 scale with 0 denoting no itch and 10, the worst itch possible. Participants were asked at 3 different time points (1 hour, 4 hours and 24 hours) after surgery to rate their itching. In the results here we reported any itching (a score greater than zero on the ItchyQuant scale) at 24 hours after surgery in each group.
Time Frame: Within first 24 hours after cesarean section
Population: Sixty-seven patients completed the protocol; of these, 34 received intramuscular promethazine (IMP) and 33 received intramuscular saline placebo (NS). There was incomplete data for 2 patients who received IMP and 1 patient who received NS.
Measure: Count of Participants; unit: Participants
Arm/Group | Promethazine | Placebo
Number analyzed (Participants) | 32 | 32
Participants
  No Itching at 24 hour | 22 | 17
  Itching at 24 hour | 10 | 15

2. Secondary Outcome: Does Promethazine Impact Level of Consciousness Compared to Placebo After Cesarean Delivery?
Description: Level of consciousness will be quantified by the RASS Scale. The RASS scale is scored with +4 to -5 scale with +4=combative, 0=alert and calm and -5=unrousable. Participants were asked at 3 different time points (1 hour, 4 hours and 24 hours) after surgery to rate their level of consciousness. In the results here we reported any score not noted to be 0 (alert and calm) at 24 hours after surgery in each group.
Time Frame: Within first 24 hours post cesarean section
Measure: Count of Participants; unit: Participants
Arm/Group | Promethazine | Placebo
Number analyzed (Participants) | 32 | 32
Participants
  Alert and Calm at 24 hour | 32 | 31
  Not Alert and Calm at 24 hour | 0 | 1

3. Secondary Outcome: Does Promethazine Change Nausea and Vomiting After Cesarean Compared to Normal Saline?
Description: We asked patients to rate their sensation of nausea and/or vomiting as none, mild, moderate or severe at 4 time points after cesarean (1 hour, 4 hours and 24 hours after cesarean). Here, we rate any report of nausea and/or vomiting as opposed to no nausea and/or vomiting at 24 hours after cesarean among the patients who had Promethazine and normal saline.
Time Frame: Within first 24 hours post cesarean section
Measure: Count of Participants; unit: Participants
Arm/Group | Promethazine | Placebo
Number analyzed (Participants) | 32 | 32
Participants
  No nausea or vomiting at 24 hours | 31 | 32
  Nausea and/or vomiting at 24 hours | 1 | 0

ADVERSE EVENTS:
Time Frame: 24 hours after study drug administration
Arm/Group | Promethazine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 0/34 | 0/33

LIMITATIONS AND CAVEATS:
We failed to enroll the planned number of patients due to a variety of factors, including challenges in availability of the study drug coupled with slow enrollment. Over two-thirds of the patients who were screened and were able to be contacted prior to surgery declined to participate. This did not support continuing enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT04805073/Prot_SAP_001.pdf